CLINICAL TRIAL: NCT01874847
Title: PLAY GAME: Post-concussion Syndrome Affecting Youth: GABAergic Effects of Melatonin. A Randomized Double-blind Placebo-controlled Trial of MELATONIN
Brief Title: PLAY GAME: Post-concussion Syndrome in Youth - Assessing the GABAergic Effects of Melatonin
Acronym: PLAYGAME
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Calgary (Other)
Collaborators: Children's Hospital of Eastern Ontario (Other)
Responsible Party: Principal Investigator, Dr. Karen Barlow, Principal Investigator, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TMT-127046
Record Dates: First submitted 2013-06-06; First posted 2013-06-11 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Post-concussion Syndrome; Post-concussive Symptoms; Traumatic Brain Injury; Concussion; Children
Keywords: melatonin; placebo; post-concussion syndrome; mild traumatic brain injury; concussion; treatment; outcome; children; functional magnetic resonance imaging; transcranial magnetic stimulation; sleep
MeSH Terms: conditions — Post-Concussion Syndrome; Brain Injuries, Traumatic; Brain Concussion | interventions — Melatonin; Sugars

STUDY DESIGN:
Intervention Model Description: Placebo controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blinded
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Melatonin 10mg (Experimental): Melatonin 10mg capsule(high dose arm), oral, once at night, given for 28 days
  Interventions: Dietary Supplement: Melatonin
- Sugar Pill (Placebo Comparator): Sugar Pill, one capsule, once at night, 28 days
  Interventions: Dietary Supplement: Sugar pill
- Melatonin 3mg (Experimental): Melatonin 3mg capsule (low dose arm), once, at night, 28 days
  Interventions: Dietary Supplement: Melatonin

INTERVENTIONS:
Dietary Supplement: Melatonin — Melatonin 10mg or 3mg capsule, one will be given at night, for 28 days
  Arms: Melatonin 10mg; Melatonin 3mg
Dietary Supplement: Sugar pill — Sugar pill will be given, one capsule, once at night, for 28 days
  Arms: Sugar Pill

SUMMARY:
PURPOSE: The long-term goal of this line of research is to develop rational, biologically based evidence for the treatment of post-concussion syndrome (PCS) in children. The objective of this application is to examine the effect of melatonin on the symptoms of PCS and its neurobiology using integrated neurodiagnostic techniques in children.

OVERVIEW: PCS is a constellation of clinical symptoms including physical (i.e. headaches), cognitive (i.e. memory), and behavioral disturbances. PCS is associated with significant morbidity in the child and his/her family), and yet there are no evidence-based medical treatments available. This suggests an urgent need to develop novel treatment options to improve outcomes for children suffering from PCS. Melatonin has several relevant mechanisms of action, and neuroprotective effects. Recent research suggests that the explanations for persistent PCS symptoms may be due to alterations in neurotransmissions and neuronal circuitry, particularly involving the dorsolateral prefrontal cortex (DLPFC). Investigators have two specific aims:

1. To determine if treatment with melatonin improves PCS in children following mild traumatic brain injury. Hypothesis: treatment of mTBI children with PCS with 3mg or 10mg of oral melatonin for 28 days will result in a decrease in PCS symptoms as compared with placebo. Effects will be dose-dependent and may be independent of sleep effects. Methods: A randomized double blind, placebo controlled trial (RCT); Outcome measure is a PCS symptom questionnaire. A subsequent RCT will then be performed using the optimal melatonin dose at a second centre.
2. To understand the neurophysiological mechanisms of paediatric PCS and assess any resultant effects of treatment with melatonin. Methods: A case-controlled study within the RCT, using functional MRI and Transcranial Magnetic Stimulation to investigate the neurophysiological properties of paediatric mTBI before and after treatment; Treatment groups from the RCT will be compared with two control groups: i) normal controls and ii) asymptomatic mTBI children.

SIGNIFICANCE: This study has the potential to 1) provide a safe and effective treatment for PCS and 2) will provide valuable information about the neurophysiological properties of the brain associated with PCS following mTBI in children and how these change with symptom resolution.

DETAILED DESCRIPTION:
We hypothesize that the treatment of children with PCS following mTBI with 3mg or 10mg of Melatonin for 28 days will result in a decrease in PCS symptoms as compared with placebo.

Primary research question:

Does the treatment of children with PCS symptoms following mTBI with 3mg sublingual Melatonin or 10mg of sublingual Melatonin for 28 days result in a decrease in PCS (physical, cognitive and behavioural) symptoms as compared with placebo?

Secondary research questions:

Is there a dose-response relationship? Is the treatment effect independent of the effect on sleep?

Research Design:

This study will be conducted as a randomized, double blind, placebo-controlled superiority trial. Three parallel treatment groups will be examined with a 1:1:1 allocation: 1) sublingual placebo, 2) sublingual Melatonin 3mg, and 3) sublingual Melatonin 10mg. Groups will be allocated using a randomization sequence that will be created in variable random block sizes (multiples of 3: 3, 6, and 9) to aid in concealment of next allocation, using random number generating software. The primary endpoint is the change on the Post-Concussion Symptom Inventory Score for parent and adolescent. The design allows for dose dependent response assessment.

Study Setting: Two academic children's hospitals in Canada Target Population: All children aged 13 to 18 years presenting to the ED of ACH and CHEO with a mTBI who remain symptomatic at 30 days post-injury.

Intervention:

Eligible patients will be randomized in equal proportions between three groups: placebo, 3mg Melatonin and 10mg Melatonin. Medication is taken sublingually one hour before sleep time at night for 28 days and will be continued even if there is symptom resolution.

Rationale for proposed dosages: Receptor-mediated effects occur at physiological doses (e.g., in children with chronic insomnia effects are achieved at 0.05-0.15mg/kg). However, to achieve non-Melatonin receptor mediated effects (e.g. GABAergic effects, direct free radical scavenging and antioxidant effects) may require supra-physiological doses. 3mg Melatonin is a standard dose used in clinical practice and lower doses do not achieve the same analgesic and anxiolytic effects; however, 3mg may be insufficient to saturate Melatonin receptors and could fall short of the supraphysiological doses we are aiming for to achieve the non-receptor mediated effects. To do this, a higher dose of 10mg will be used which is a logarithmical increase and is still in a clinically acceptable range.

Modifications: No serious side effects have been reported with Melatonin treatment at the above doses. Higher doses (70mg/day) have been used in children with muscular dystrophy with no adverse events. Occasionally excessive daytime sleepiness has been reported which should be reported as an adverse event. This usually resolves in a few days. Treatment should continue unless the sleepiness is problematic for more than 3 days in which case half a tablet may be tried (after reporting this to the study team).

Adherence:

Administration of study pill will occur at home under the supervision of the parent. When the study pill is dispensed, the research coordinator will review the importance of following study guidelines, instructions about taking study pills including timing, storage, and what to do in the event of a missed dose. Instructions about the purpose, use, and care of the study pill will be included with the package. Families will be notified that there will be a pill count at every study visit and the importance of calling the clinic if experiencing problems possibly related to study product such as symptoms, or lost pills. Methodologies to maximize follow-up and compliance include convenient follow-up times, participant engagement strategies (e.g. newsletters, website) and experienced research personnel.

Adherence assessments will include a daily diary, and abreview of the medication log, pill count every week, and a review of reasons for non-compliance. Unused tablets will be counted and recorded on the appropriate case report form.

Concomitant care: There are no restrictions on the use of other medications. All participants will be advised to try to avoid analgesia overuse. Participants will be asked to complete a diary of any medications, medical appointments and alternative therapies.

ELIGIBILITY:
Inclusion Criteria:

* Concussion/mild traumatic brain injury trauma with an increase in symptoms (increase in PCS symptoms compared with pre-injury status) at 30 days post injury
* must be able to swallow pills

Exclusion Criteria:

* Previous significant medical history, or previous concussion within 3 months
* Participant in a natural history study of concussion
* Lactose intolerance, as the placebo contains lactose
* Use of drugs that are likely to affect TMS, fMRI and/or sleep
* Inability to complete questionnaires/evaluation e.g. non-English language

Ages: 8 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 99 (Actual)
Dates: Start 2013-09; Primary Completion 2017-04 (Actual); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Change on the Post Concussion Symptom Inventory (PCSI)-(8 - 18 years) | Baseline, 4 weeks and 12 weeks
  The PCSI is a standardized questionnaire of 26 symptoms provides an overall rating of Post concussion symptoms. It has four specific domains: physical (including headaches), cognitive, emotional (including mood) and fatigue and high level of internal consistency, alpha=0.92. Parent and youth PCSI scores correlate. Low symptom rates are found in normative samples. The version for youth will also be recorded (PCSI-Y). Change in PCSI scores allows us to account for baseline variability and gender.

SECONDARY OUTCOMES:
Number of Patient's Adverse Events | 1, 2, 3 and 4 weeks

OTHER OUTCOMES:
Change on the Child Health Questionnaire (CHQ) | Baseline, 4 and 12 weeks
  Parent and child rating of functional impairment will be obtained using the 50-item Child Health Questionnaire, parent CHQ-Parent Form (PF)50 and child, CHQ-Child Form (CF)87. The reliability and validity is established in TBI and PCS.
Change on the Behavior Assessment System for Children (BASC)-2 -Parent | Baseline, 4 and 12 weeks
  BASC-2 is a standardized parent report measure of child behavior consisting of 150 items. It provides an indication of internalizing and externalizing behaviour (e.g., anxiety, depression). Items are rated using true-false, or a 4-point ordinal scale.
  The internal consistency for the composite subscales range from .87 to .96 and test-retest reliability is high, ranging from .81 to .96 (10-20 minutes) (
Change on the Post Concussion Symptom Inventory (PCSI)- Parent questionnaire | Baseline, 2 , 4 and 12 weeks
  The PCSI is a standardized questionnaire of 26 symptoms provides an overall rating of Post concussion symptoms. It has four specific domains: physical (including headaches), cognitive, emotional (including mood) and fatigue and high level of internal consistency, alpha=0.92. Parent and youth PCSI scores correlate. Low symptom rates are found in normative samples. The version for youth will also be recorded (PCSI-Y). Change in PCSI scores allows us to account for baseline variability and gender.

CONTACTS AND LOCATIONS:
Overall Officials: Karen M Barlow, MB.ChB, Principal Investigator — Alberta Children's Hospital Research Institute, University of Calgary
Locations (1):
- Alberta Children's Hospital, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD

REFERENCES:
- [Background] Kuczynski A, Crawford S, Bodell L, Dewey D, Barlow KM. Characteristics of post-traumatic headaches in children following mild traumatic brain injury and their response to treatment: a prospective cohort. Dev Med Child Neurol. 2013 Jul;55(7):636-41. doi: 10.1111/dmcn.12152. Epub 2013 Apr 5. PMID 23560811
- [Background] Barlow KM, Crawford S, Stevenson A, Sandhu SS, Belanger F, Dewey D. Epidemiology of postconcussion syndrome in pediatric mild traumatic brain injury. Pediatrics. 2010 Aug;126(2):e374-81. doi: 10.1542/peds.2009-0925. Epub 2010 Jul 26. PMID 20660554
- [Background] Barlow KM, Brooks BL, MacMaster FP, Kirton A, Seeger T, Esser M, Crawford S, Nettel-Aguirre A, Zemek R, Angelo M, Kirk V, Emery CA, Johnson D, Hill MD, Buchhalter J, Turley B, Richer L, Platt R, Hutchison J, Dewey D. A double-blind, placebo-controlled intervention trial of 3 and 10 mg sublingual melatonin for post-concussion syndrome in youths (PLAYGAME): study protocol for a randomized controlled trial. Trials. 2014 Jul 7;15:271. doi: 10.1186/1745-6215-15-271. PMID 25001947
- [Derived] Iyer KK, Zalesky A, Cocchi L, Barlow KM. Neural Correlates of Sleep Recovery following Melatonin Treatment for Pediatric Concussion: A Randomized Controlled Trial. J Neurotrauma. 2020 Dec 15;37(24):2647-2655. doi: 10.1089/neu.2020.7200. Epub 2020 Sep 14. PMID 32772826
- [Derived] Barlow KM, Brooks BL, Esser MJ, Kirton A, Mikrogianakis A, Zemek RL, MacMaster FP, Nettel-Aguirre A, Yeates KO, Kirk V, Hutchison JS, Crawford S, Turley B, Cameron C, Hill MD, Samuel T, Buchhalter J, Richer L, Platt R, Boyd R, Dewey D. Efficacy of Melatonin in Children With Postconcussive Symptoms: A Randomized Clinical Trial. Pediatrics. 2020 Apr;145(4):e20192812. doi: 10.1542/peds.2019-2812. Epub 2020 Mar 26. PMID 32217739
- See also: PlayGame Trial website — http://www.playgametrial.ca